CLINICAL TRIAL: NCT03699358
Title: Does Myeloid or Lymphoid Origin of Hematologic Neoplasm Affect Pulmonary Functions, Muscle Strength, Exercise Capacity, Fatigue and Quality of Life?
Brief Title: Physical Impairments Related to Myeloid and Lymphoid Malignancies
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Other Study IDs: GaziUniversity15
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Stem Cell Transplantation
Keywords: hematopoietic stem cell transplantation; respiratory function test; respiratory muscles; muscle strength; exercise; walk test; quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Myeloid recipients: Patients diagnosed with hematologic malignancy were recipients who undergone allogeneic-HSCT. Recipients were included in the current study and grouped as myeloid and lymphoid according to origin of their diagnosis. Recipients who had myeloid type disorders were included in myeloid group as well as recipients who had lymphoid type disorders were included in lymphoid group.
- Group 2: Lymphoid recipients: Patients diagnosed with hematologic malignancy were recipients who undergone allogeneic-HSCT. Recipients were included in the current study and grouped as myeloid and lymphoid according to origin of their diagnosis. Recipients who had myeloid type disorders were included in myeloid group as well as recipients who had lymphoid type disorders were included in lymphoid group.

SUMMARY:
Hematologic malignancies may arise from myeloid and lymphoid blood cells lineages affecting blood, bone marrow and lymph nodes. Accordingly, negative effects of malignancies on body systems vary. As known, muscle strength, exercise capacity, fatigue and quality of life deteriorate during allogeneic hematopoietic stem cell transplantation (HSCT). However, impacts of myeloid and lymphoid type disorders on pulmonary functions, muscle strength, exercise capacity, fatigue and quality of life in allogeneic-HSCT who diagnosed with hematologic malignancies. Therefore, current study aimed to comparatively investigate physical impairments between recipients with hematologic malignancies according to myeloid and lymphoid type disorder.

DETAILED DESCRIPTION:
Hematologic malignancies affecting blood, bone marrow and lymph nodes comprise neoplasm of either myeloid or lymphoid blood stem cells origin. While a lymphoid stem cell becomes a white blood cell, a myeloid stem cell becomes one of the red blood cells, white blood cells or platelets types. Due to the this reason, defects in myeloid stem cells result in acute and chronic myelogenous leukemia, myelodysplastic syndromes or myeloproliferative diseases, whereas defects in lymphoid stem cells result in lymphomas, lymphocytic leukemias or myeloma. On the other hand, most of these hematologic malignancies are characterized with high rate of morbidity and mortality because of both the nature and various toxic treatments of neoplasm including chemotherapy with multiple agents, corticosteroids and hematopoietic stem cell transplantation (HSCT). Especially after allogeneic-HSCT, recipients experience more impairments in pulmonary functions, respiratory and peripheral muscle strength, exercise capacity, perception of fatigue and quality of life scores which make their lives difficult in terms of actively trying to return to the their life. However, although it has been known that each hematologic disease has a different negative impact on varied body systems or organs after HSCT, little attention has been paid to the comparatively investigation of impacts of myeloid and lymphoid hematological malignancies on pulmonary functions, muscle strength, exercise capacity, fatigue and quality of life in allogeneic-HSCT recipients. Hence, current study aimed to comparatively investigate physical impairments between recipients with hematologic malignancies according to myeloid and lymphoid type disorder.

Recipients undergone allogeneic-HSCT (˃100 days post-HSCT status) were included. Hematologic malignancies were grouped as myeloid and lymphoid. Pulmonary functions (spirometry), peripheral (dynamometer) and respiratory muscle strength (MIP-MEP) (mouth pressure device), exercise capacity (Modified Incremental Shuttle Walk Test (ISWT)), and quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age,
* being an allogeneic-HSCT recipient who was at minimum 100 days status after transplantation
* receiving optimal standard medical therapy including immunosuppressive agents, antibiotics, supplements and other drugs.

Exclusion Criteria:

* having cognitive disorders, orthopedic or neurological disease with a potential to affect assessment of exercise capacity, visual impairments and mucositis which may prevent measurements, comorbidities such as asthma, chronic obstructive pulmonary disease (COPD), acute respiratory or other infections, acute hemorrhage, low hemoglobin values (≤8 g/L) and low platelet count (≤10.000 mm3).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in Bone Marrow Transplantation Unit of University were referred for participation in rehabilitation program as outpatient to Faculty of Health Science of University, Department of Physiotherapy and Rehabilitation, cardiopulmonary rehabilitation unit. Patients diagnosed with hematologic malignancy were recipients who undergone allogeneic-HSCT. Recipients who had myeloid type disorders were included in myeloid group as well as recipients who had lymphoid type disorders were included in lymphoid group. A physiotherapist conducted all measurements in the same day for all recipients individually.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Maximal exercise capacity evaluation | 15-20 minutes
  Modified-Incremental Shuttle Walk Test (ISWT) test was used to evaluate maximal exercise capaciity.

SECONDARY OUTCOMES:
pulmonary function test | 5 minutes
  This test was evaluated using a spirometry
Inspiratory and expiratory muscle strength (MIP, MEP) | 5-10 minutes
  Respiratory muscle strength was evaluated with a mouth pressure device
Quadriceps femoris muscle strength | 5 minutes
  Peripheral muscle strength was evaluated with a hand-held dynamometer
Quality of life level | 2 minutes
  The Turkish version of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version3.0 (EORTC QLQ-C30) was carried out to the recipients for evaluation of aspects of quality of life impairment which is a valid and reliable questionnaire for patients with cancer in the whole world.Self-administered questionnaire incorporates five functional scales including social functioning subscale, three symptom scales including fatigue subscale, and a global health status as well as several single items. All item scores are transformed to percents (0-100). Higher values represent higher functional/healthy level in functional scales, a higher quality of life level in global health status and increased presence of symptoms in symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, PhD, Study Chair — Gazi University; Meral Boşnak Güçlü, PhD, Study Director — Gazi University; Gülsan Türköz Sucak, PhD., Principal Investigator — Bahçeşehir University
Locations (1):
- Gazi University Faculty of Health Science Department of PhysioTherapy, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- [Background] Paul KL. Rehabilitation and exercise considerations in hematologic malignancies. Am J Phys Med Rehabil. 2011 May;90(5 Suppl 1):S88-94. doi: 10.1097/PHM.0b013e31820be055. PMID 21765268
- [Background] Bergenthal N, Will A, Streckmann F, Wolkewitz KD, Monsef I, Engert A, Elter T, Skoetz N. Aerobic physical exercise for adult patients with haematological malignancies. Cochrane Database Syst Rev. 2014 Nov 11;(11):CD009075. doi: 10.1002/14651858.CD009075.pub2. PMID 25386666
- [Background] Steinberg A, Asher A, Bailey C, Fu JB. The role of physical rehabilitation in stem cell transplantation patients. Support Care Cancer. 2015 Aug;23(8):2447-60. doi: 10.1007/s00520-015-2744-3. Epub 2015 May 14. PMID 25971213
- [Background] Bargi G, Bosnak Guclu M, Turkoz Sucak AG. Differences in pulmonary and extra-pulmonary characteristics in severely versus non-severely fatigued recipients of allogeneic hematopoietic stem cell transplantation: a cross-sectional, comparative study. Hematology. 2019 Dec;24(1):112-122. doi: 10.1080/10245332.2018.1526441. Epub 2018 Sep 27. PMID 30261831